CLINICAL TRIAL: NCT04434924
Title: The Construction of Precision Medicine in Chinese Medicine
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH109-REC1-025
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hypertension
Keywords: Traditional Chinese precision medicine; Chinese medicine immunoassay; Body constitution; genetic variation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"Precise medicine" is also called "personal medicine". With the development of big data database, genetic testing and artificial intelligence, the concept of precision medicine has been applied to the diagnosis, treatment and prevention of different diseases. Traditional Chinese medicine (TCM) has traditionally emphasis on personalized medicine, according to each person's body constitution, through discriminatory treatment and personalized treatment methods. Chinese medicine doctors collect patients' information to distinguish the type of TCM pattern, and then according to the different types of diagnosis of traditional Chinese medicine to decide of using herbs, acupuncture, massage and other treatment strategies. However, lacking of objective data of traditional Chinese medicine, the current research on precision medicine in Chinese medicine is still limited. The aim of this study is to establish a big database of traditional Chinese precision medicine, and use the patients with hypertension as the population to conduct research on precision medicine in Chinese medicine.This study will combine the TCM body constitutional questionnaire, tongue diagnosis, pulse diagnosis, Chinese medicine immunoassay and genetic testing. In addition, the information providing by the medical electronic medical record system of China Medical University Hospital will be connected, which include modern medical diagnosis, treatment, blood and biochemical analysis and imaging. We will combine the big data analysis and artificial intelligence interpretation technology to explore the correlation between different TCM syndrome types and gene variations in patients with hypertension and establish a database of TCM precision medicine. We will also conduct the education training and symposium to train TCM precision medical talents and promote public understanding of TCM precision medicine. This project will establish a database of traditional Chinese medicine precision medicine to provide the correlation between different TCM pattern types of patients with hypertension, the reaction to different herbal medicine, and gene mutation, and provide reference for TCM clinicians.

ELIGIBILITY:
Inclusion Criteria:

1. Primary hypertension
2. Older than 20 year-old

Exclusion Criteria:

1. Past history of cancer
2. Hemodialysis
3. Hypertension caused by renal diseases or endocrine disorders
4. Pregnancy
5. Patients can not received investigation of body constitution, TCM tongue examination and pulse examination

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed as having primary hypertension by cardiologists.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
The correlation between TCM body constitution and genetic variation | 2 years
  The correlation between TCM body constitution and genetic variation of patients with primary hypertension will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan